CLINICAL TRIAL: NCT04350398
Title: Effect of Multidisciplinary Management by Hippotherapy on the Quality of Life of Women With a Diagnosis of Breast Cancer: Randomized Controlled Clinical Trial on the Effectiveness of the Therapeutic Intervention
Brief Title: Rehabilitation Through Hippotherapy for the Management of Women After Primary Treatment of Breast Cancer
Acronym: HippoBreastCa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance Equiphoria (Other)
Collaborators: Institut Equiphoria - La Canourgue, France (Unknown); Montpellier Institut du Sein - Montpellier, France (Unknown); Clinique Clementville - Montpellier, France (Unknown); Klésia Languedoc Service de l'Action Sociale - France (Unknown); Fondation Crédit Agricole Solidarité et Développement - France (Unknown); Crédit Agricole du Languedoc - France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-A01656-45
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Female; Side Effects; Psychological Distress; Physical Disability
Keywords: Breast cancer; Hippotherapy; Global rehabilitation; Quality of life; Body image; Cognitive impairment; Fatigue; Anxiety and depression; Physical impairment; Psychological reinforcement; Social reintegration
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Fatigue; Anxiety Disorders; Depression | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: A randomized simple-blind controlled trial on efficacy of the hippotherapy treatment against conventional one will be conducted. Patients selected will be randomly divided into 2 groups: hippotherapy treated group versus control group. To ensure that patients in the 2 groups are similar in all respects, except for the planned intervention, the randomization will be stratified by age representing respectively two stages: 1) Pre-menopause; 2) Post-menopause; and by type of treatment: A) Single treatment: surgery or chemotherapy or hormone therapy or radiotherapy; B) Two or more treatments.
Who Masked: Investigator
Masking Description: Data will be collected on the Montpellier Institut du Sein site by relying on the CRA who will follow up and check the information in due time of the self-questionnaires. The data will be duly anonymized and handled blindly. Data will be centralized on a secure server at the Equiphoria Institute. Their processing and analysis will be carried out blindly by the PI or by a private service provider (Biostatem France)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hippotherapy treated group (Experimental): During the initial week of intervention, sessions will be mainly carried on horseback. We will use the movement of the horse: (i) to allow patient re-appropriating her body and find harmony; (ii) to initiate rehabilitation of movements (shoulder, neck, upper extremity, whole body), gesture and femininity. The goal is to reconstruct a harmonic body image both in the private and public sphere, through different techniques. A few walking sessions may be needed to reinforce some landmarks.
  During the short stages the work will be mainly done by walking alongside the horse. These reinforcement periods act like a trampoline, necessary to have a new momentum providing the opportunity to take a step back from the everyday, to regenerate somehow. The reaction time is generally optimized considering the imprint done during the initial long stage. One of the main themes that come up during this period is fear (relapse, the future, not achieving the goals, pain, relationship issues, etc.).
  Interventions: Other: Hippotherapy
- Conventional therapy treated group (Placebo Comparator): Patients in the control group are followed by dedicated personnel of the Montpellier Institut du Sein. This personalized care pathway after/during the cancer treatment takes into consideration all aspects of the disease, allowing to coordinate the intervention of the professionals that the patient might need in order to better preserve her quality of life while answering questions about cancer, prevention, treatments, or life after illness. The MIS mobilizes a chain of skills and support by providing patients: radiologists, pathologists, surgeons, oncologists, and radiation therapists, nuclear doctors, physiotherapists, cardiologists, psychologists, psychiatrists, nurses, social workers, nutritionists, dieticians, onco-geneticists, osteopaths, homeopaths, acupuncturists, sexologists, addictologists, algologists, and vascular physicians.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Hippotherapy — The horse is an excellent collaborator in situations of physical and mental disability, whether temporary or consolidated. It provides support to humans towards an impairment (anatomical or physiological), a disability, or a restriction of participation as defined by the WHO in 2001. Hippotherapy has a direct action on the sensorimotor capacities of the individual but also on their cognitive capacities, such as attention, memory, psychomotricity, emotions, perceptions, the sequencing of complex movements, or the experience of oneself and the functions of time. Overall, the strong demand from the sensitive, sensory and motor spheres promotes and interacts with the mechanisms linked to the execution of tasks in the cognitive domain (memory, attention, executive functions, speed of information processing, etc.) through the interactions of several neural networks.
  Arms: Hippotherapy treated group
Other: Conventional therapy — Personalized care pathway after/during the cancer treatment takes into consideration all aspects of the disease, allowing to coordinate the intervention of the professionals that the patient might need in order to better preserve her quality of life while answering questions about cancer, prevention, treatments, or life after illness. The MIS mobilizes a chain of skills and support by providing patients: radiologists, pathologists, surgeons, oncologists, and radiation therapists, nuclear doctors, physiotherapists, cardiologists, psychologists, psychiatrists, nurses, social workers, nutritionists, dieticians, onco-geneticists, osteopaths, homeopaths, acupuncturists, sexologists, addictologists, algologists, and vascular physicians.
  Arms: Conventional therapy treated group

SUMMARY:
Breast cancer is the most common women's cancer and the third leading cause of death. Advances in prevention, detection and primary treatment have improved overall survival leading to its growing acceptance as a long-term disease. Following the announcement of breast cancer, but also after primary treatment, some symptoms appear directly compromising psychic and physical spheres. Hippotherapy is an emerging specialized rehabilitation approach performed through specially trained horses by accredited health professionals. The proposed hippotherapy program offers key elements for physical, psychic and social reinforcement, complementing conventional care. The aim is to provide patients with tools to consolidate their self-awareness and thus strengthen their ability to cope with the disease.

DETAILED DESCRIPTION:
Following the announcement and evolution of breast cancer, but also in response to primary treatment, some symptoms appear to directly compromise the psychic and/or physical sphere of the individual. Current rehabilitation programs are not sufficiently oriented to solve most of these symptoms. Hippotherapy is an emerging specialized rehabilitation approach, performed on a specially trained horse by accredited health professionals (e.g. medical doctors, physical therapists, occupational therapists, psychomotricians, speech-language pathologists, clinical psychologists). The horse is an excellent collaborator in situations of physical and psychic disability, whether temporary or consolidated. It provides human support for impairments (anatomical or physiological), activity limitations, and participation restrictions as defined by WHO. Hippotherapy has a direct action on the sensorimotor capacities of the individual but also on his cognitive abilities, i.e. attention, memory, psychomotricity, emotion, perception, sequencing of complex movements, self-experience, psychic temporality. Overall, the strong solicitation of the sensory and motor spheres promotes and interacts with the mechanisms related to the execution of tasks in the cognitive domain through the interactions of several neural networks. A randomized simple-blinded controlled trial on hippotherapy versus conventional care will be carried out. After giving their informed consent, patients will be enrolled in the trial. The 6-months program includes 1-week daily sessions of hippotherapy by the end of the initial cancer treatment followed by three short 2-days sessions with an interval of 2 months between each. The study will focus on 86 patients. Recruitment will be done over a 48-months' period. A battery of self-administered questionnaires will allow to study both the functional and psychological outcome. The primary end point will be quality of life, whereas body image, fatigue, anxiety, depression and cognitive performances will be the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of breast cancer staging [T1-T3, N0-N2 and M0]
* Patient already scheduled or ongoing treatment for surgery and/or chemotherapy and/or hormone therapy and/or radiotherapy
* Having consulted a physician of the Care and Support Unit of the MIS during its health care
* WHO performance index from 0 to 2
* Able to give her informed consent in writing
* Able to complete questionnaires
* Abduction of the hip necessary and sufficient (to allow horse riding)
* Affiliated to a social security scheme
* Certificate of no contraindication issued by the physician in charge

Exclusion Criteria:

* History of malignant tumors in the last 5 years with the exception of basocellular skin carcinoma or squamous cell carcinoma
* Breast cancer as a secondary diagnosis
* Medication intake or presence of conditions associated with fatigue (e.g. chronic fatigue syndrome)
* Concomitant and uncontrolled severe degenerative or chronic disease
* History of allergic reactions to dust and/or horsehair, or asthma
* Contraindications to physical activity
* History of horseback riding or hippotherapeutic treatment during the last 6 months
* Clinically significant cognitive impairment or dementia
* Pregnancy and breastfeeding
* Majors protected by law
* Patient participating in another biomedical research or in exclusion period

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life through EORTC QLQ-C30 | Before the beginning of the protocol; after the first 1-week session; at the end of the last session at 6 months
  This questionnaire was designed to be cancer specific, multidimensional in structure, suitable for self-administration (brief and easy to complete), and applicable in a wide range of cultural contexts. The scores ranges from 0 to 100, a higher score represents a higher ("better") level of functioning.

SECONDARY OUTCOMES:
Changes in Body image representation through Body Image Scale (BIS) | Before the beginning of the protocol; after the first 1-week session; at the end of the last session at 6 months
  The questionnaire focuses on patients' emotional and behavioral experiences of their body image, resulting from cancer and treatment, including aspects of perceived physical appearance, body integrity, and seduction capacity. The total score ranges from 0 to 30. A higher score means a higher level of body image disturbance.
Changes in Fatigue sensation through Multidimensional Fatigue Inventory (MFI-20) | Before the beginning of the protocol; after the first 1-week session; at the end of the last session at 6 months
  MFI seems to be one of the best questionnaires to provide a fatigue profile. Its psychometric properties have been studied in different populations and it is easy to administer. Score ranges from 0 to 100. Higher total scores correspond with more acute levels of fatigue.
Changes in anxiety and depression through Hospital Anxiety and Depression Scale (HADS) | Before the beginning of the protocol; after the first 1-week session; at the end of the last session at 6 months
  This scale was constructed excluding any item concerning somatic aspects, aspects that could be confused between physical and mental illness. It is a self-questionnaire to be completed according to oneself condition during the past week. Score ranges from 0 to 21 for each item. Higher total scores correspond to presence of the respective state.
Changes in the Cognitive sphere assessment through Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | Before the beginning of the protocol; after the first 1-week session; at the end of the last session at 6 months
  The questions are grouped into six cognitive domains (memory, verbal fluency, concentration, mental sharpness, resistance to interference, multitasking ability) and two sub-criteria (visibility of the disorder by the entourage, impact on the quality of life). 37-item ranging from 0 to 4 consist of four subscales. Higher scores represent better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Gaviria, MD, PhD, Study Director — Alliance Equiphoria
Locations (1):
- Institut Equiphoria, La Canourgue, France

IPD SHARING:
Plan to Share IPD: Undecided
Dissemination of study results will be done through a classic strategy for publications (reports, scientific publications) and communications (congresses, meetings). The coordinator will be in charge of the dissemination strategy. Controlled access to the final trial dataset will be given when a reasonable request has a precise and valid scientific aim. Thus, we will protect the rights of patients and the intellectual property of the scientists who designed the trial and collected the data.

REFERENCES:
- [Background] Khan F, Amatya B, Ng L, Demetrios M, Zhang NY, Turner-Stokes L. Multidisciplinary rehabilitation for follow-up of women treated for breast cancer. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD009553. doi: 10.1002/14651858.CD009553.pub2. PMID 23235677
- [Background] Hulka BS, Moorman PG. Breast cancer: hormones and other risk factors. Maturitas. 2001 Feb 28;38(1):103-13; discussion 113-6. doi: 10.1016/s0378-5122(00)00196-1. PMID 11311599
- [Background] Belot A, Grosclaude P, Bossard N, Jougla E, Benhamou E, Delafosse P, Guizard AV, Molinie F, Danzon A, Bara S, Bouvier AM, Tretarre B, Binder-Foucard F, Colonna M, Daubisse L, Hedelin G, Launoy G, Le Stang N, Maynadie M, Monnereau A, Troussard X, Faivre J, Collignon A, Janoray I, Arveux P, Buemi A, Raverdy N, Schvartz C, Bovet M, Cherie-Challine L, Esteve J, Remontet L, Velten M. Cancer incidence and mortality in France over the period 1980-2005. Rev Epidemiol Sante Publique. 2008 Jun;56(3):159-175. doi: 10.1016/j.respe.2008.03.117. Epub 2008 Jun 10. PMID 18547762
- [Background] Klein D, Mercier M, Abeilard E, Puyraveau M, Danzon A, Dalstein V, Pozet A, Guizard AV, Henry-Amar M, Velten M. Long-term quality of life after breast cancer: a French registry-based controlled study. Breast Cancer Res Treat. 2011 Aug;129(1):125-34. doi: 10.1007/s10549-011-1408-3. Epub 2011 Feb 22. PMID 21340477
- [Background] Miaskowski C, Dibble SL. The problem of pain in outpatients with breast cancer. Oncol Nurs Forum. 1995 Jun;22(5):791-7. PMID 7675686
- [Background] Hopwood P, Haviland JS, Sumo G, Mills J, Bliss JM, Yarnold JR; START Trial Management Group. Comparison of patient-reported breast, arm, and shoulder symptoms and body image after radiotherapy for early breast cancer: 5-year follow-up in the randomised Standardisation of Breast Radiotherapy (START) trials. Lancet Oncol. 2010 Mar;11(3):231-40. doi: 10.1016/S1470-2045(09)70382-1. Epub 2010 Feb 6. PMID 20138809
- [Background] Lauridsen MC, Christiansen P, Hessov I. The effect of physiotherapy on shoulder function in patients surgically treated for breast cancer: a randomized study. Acta Oncol. 2005;44(5):449-57. doi: 10.1080/02841860510029905. PMID 16118078
- [Background] Howard-Anderson J, Ganz PA, Bower JE, Stanton AL. Quality of life, fertility concerns, and behavioral health outcomes in younger breast cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Mar 7;104(5):386-405. doi: 10.1093/jnci/djr541. Epub 2012 Jan 23. PMID 22271773
- [Background] Demark-Wahnefried W, Winer EP, Rimer BK. Why women gain weight with adjuvant chemotherapy for breast cancer. J Clin Oncol. 1993 Jul;11(7):1418-29. doi: 10.1200/JCO.1993.11.7.1418. PMID 8315439
- [Background] Lee JJ, Swain SM. Peripheral neuropathy induced by microtubule-stabilizing agents. J Clin Oncol. 2006 Apr 1;24(10):1633-42. doi: 10.1200/JCO.2005.04.0543. PMID 16575015
- [Background] Burgess C, Cornelius V, Love S, Graham J, Richards M, Ramirez A. Depression and anxiety in women with early breast cancer: five year observational cohort study. BMJ. 2005 Mar 26;330(7493):702. doi: 10.1136/bmj.38343.670868.D3. Epub 2005 Feb 4. PMID 15695497
- [Background] Christensen S, Zachariae R, Jensen AB, Vaeth M, Moller S, Ravnsbaek J, von der Maase H. Prevalence and risk of depressive symptoms 3-4 months post-surgery in a nationwide cohort study of Danish women treated for early stage breast-cancer. Breast Cancer Res Treat. 2009 Jan;113(2):339-55. doi: 10.1007/s10549-008-9920-9. Epub 2008 Feb 16. PMID 18278553
- [Background] Galiano-Castillo N, Ariza-Garcia A, Cantarero-Villanueva I, Fernandez-Lao C, Diaz-Rodriguez L, Arroyo-Morales M. Depressed mood in breast cancer survivors: associations with physical activity, cancer-related fatigue, quality of life, and fitness level. Eur J Oncol Nurs. 2014 Apr;18(2):206-10. doi: 10.1016/j.ejon.2013.10.008. Epub 2013 Nov 5. PMID 24201014
- [Background] Mehnert A, Berg P, Henrich G, Herschbach P. Fear of cancer progression and cancer-related intrusive cognitions in breast cancer survivors. Psychooncology. 2009 Dec;18(12):1273-80. doi: 10.1002/pon.1481. PMID 19267364
- [Background] van Dam FS, Schagen SB, Muller MJ, Boogerd W, vd Wall E, Droogleever Fortuyn ME, Rodenhuis S. Impairment of cognitive function in women receiving adjuvant treatment for high-risk breast cancer: high-dose versus standard-dose chemotherapy. J Natl Cancer Inst. 1998 Feb 4;90(3):210-8. doi: 10.1093/jnci/90.3.210. PMID 9462678
- [Background] Schagen SB, Muller MJ, Boogerd W, Rosenbrand RM, van Rhijn D, Rodenhuis S, van Dam FS. Late effects of adjuvant chemotherapy on cognitive function: a follow-up study in breast cancer patients. Ann Oncol. 2002 Sep;13(9):1387-97. doi: 10.1093/annonc/mdf241. PMID 12196364
- [Background] Fan HG, Houede-Tchen N, Yi QL, Chemerynsky I, Downie FP, Sabate K, Tannock IF. Fatigue, menopausal symptoms, and cognitive function in women after adjuvant chemotherapy for breast cancer: 1- and 2-year follow-up of a prospective controlled study. J Clin Oncol. 2005 Nov 1;23(31):8025-32. doi: 10.1200/JCO.2005.01.6550. PMID 16258100
- [Background] Myers JS. Chemotherapy-related cognitive impairment: the breast cancer experience. Oncol Nurs Forum. 2012 Jan;39(1):E31-40. doi: 10.1188/12.ONF.E31-E40. PMID 22201666
- [Background] Reid-Arndt SA, Hsieh C, Perry MC. Neuropsychological functioning and quality of life during the first year after completing chemotherapy for breast cancer. Psychooncology. 2010 May;19(5):535-44. doi: 10.1002/pon.1581. PMID 19472296
- [Background] Gokal K, Munir F, Wallis D, Ahmed S, Boiangiu I, Kancherla K. Can physical activity help to maintain cognitive functioning and psychosocial well-being among breast cancer patients treated with chemotherapy? A randomised controlled trial: study protocol. BMC Public Health. 2015 Apr 23;15:414. doi: 10.1186/s12889-015-1751-0. PMID 25903195
- [Background] Bloom JR, Stewart SL, Chang S, Banks PJ. Then and now: quality of life of young breast cancer survivors. Psychooncology. 2004 Mar;13(3):147-60. doi: 10.1002/pon.794. PMID 15022150
- [Background] Gilbert E, Ussher JM, Perz J. Sexuality after breast cancer: a review. Maturitas. 2010 Aug;66(4):397-407. doi: 10.1016/j.maturitas.2010.03.027. Epub 2010 May 2. PMID 20439140
- [Background] Hoving JL, Broekhuizen ML, Frings-Dresen MH. Return to work of breast cancer survivors: a systematic review of intervention studies. BMC Cancer. 2009 Apr 21;9:117. doi: 10.1186/1471-2407-9-117. PMID 19383123
- [Background] Islam T, Dahlui M, Majid HA, Nahar AM, Mohd Taib NA, Su TT; MyBCC study group. Factors associated with return to work of breast cancer survivors: a systematic review. BMC Public Health. 2014;14 Suppl 3(Suppl 3):S8. doi: 10.1186/1471-2458-14-S3-S8. Epub 2014 Nov 24. PMID 25437351
- [Background] Ganz PA, Rowland JH, Desmond K, Meyerowitz BE, Wyatt GE. Life after breast cancer: understanding women's health-related quality of life and sexual functioning. J Clin Oncol. 1998 Feb;16(2):501-14. doi: 10.1200/JCO.1998.16.2.501. PMID 9469334
- [Background] Tiggemann M. Body image across the adult life span: stability and change. Body Image. 2004 Jan;1(1):29-41. doi: 10.1016/S1740-1445(03)00002-0. PMID 18089139
- [Background] Baucom DH, Porter LS, Kirby JS, Gremore TM, Keefe FJ. Psychosocial issues confronting young women with breast cancer. Breast Dis. 2005-2006;23:103-13. doi: 10.3233/bd-2006-23114. PMID 16823173
- [Background] Rooney M, Wald A. Interventions for the management of weight and body composition changes in women with breast cancer. Clin J Oncol Nurs. 2007 Feb;11(1):41-52. doi: 10.1188/07.CJON.41-52. PMID 17441396
- [Background] Perry S, Kowalski TL, Chang CH. Quality of life assessment in women with breast cancer: benefits, acceptability and utilization. Health Qual Life Outcomes. 2007 May 2;5:24. doi: 10.1186/1477-7525-5-24. PMID 17474993
- [Background] Masini A. Equine-assisted psychotherapy in clinical practice. J Psychosoc Nurs Ment Health Serv. 2010 Oct;48(10):30-4. doi: 10.3928/02793695-20100831-08. Epub 2010 Sep 22. PMID 20873699
- [Background] Cerulli C, Minganti C, De Santis C, Tranchita E, Quaranta F, Parisi A. Therapeutic horseback riding in breast cancer survivors: a pilot study. J Altern Complement Med. 2014 Aug;20(8):623-9. doi: 10.1089/acm.2014.0061. Epub 2014 Jun 25. PMID 24963599
- [Background] Costa DS, Aaronson NK, Fayers PM, Pallant JF, Velikova G, King MT. Testing the measurement invariance of the EORTC QLQ-C30 across primary cancer sites using multi-group confirmatory factor analysis. Qual Life Res. 2015 Jan;24(1):125-33. doi: 10.1007/s11136-014-0799-0. Epub 2014 Sep 6. PMID 25193618
- [Background] Joly F, Lange M, Rigal O, Correia H, Giffard B, Beaumont JL, Clisant S, Wagner L. French version of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) version 3. Support Care Cancer. 2012 Dec;20(12):3297-305. doi: 10.1007/s00520-012-1439-2. Epub 2012 May 2. PMID 22549504
- [Background] Smets EM, Garssen B, Cull A, de Haes JC. Application of the multidimensional fatigue inventory (MFI-20) in cancer patients receiving radiotherapy. Br J Cancer. 1996 Jan;73(2):241-5. doi: 10.1038/bjc.1996.42. PMID 8546913
- [Background] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145
- [Derived] Viruega H, Galy C, Loriette C, Jacquot S, Houpeau JL, Gaviria M. Breast Cancer: How Hippotherapy Bridges the Gap between Healing and Recovery-A Randomized Controlled Clinical Trial. Cancers (Basel). 2023 Feb 19;15(4):1317. doi: 10.3390/cancers15041317. PMID 36831658